CLINICAL TRIAL: NCT02577497
Title: Effect of Extra- Fine Versus Coarse-Particle Inhaled Corticosteroids (ICS) on Ventilation Heterogeneity in Children With Poorly Controlled Asthma
Acronym: EXPAND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Willliam Gerald Teague, Chief, Division of Respiratory Medicine, Allergy, and Immunology, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 18422
Record Dates: First submitted 2015-10-08; First posted 2015-10-16 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Fluticasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Beclomethasone (Experimental): Subjects are being randomized to 8 weeks of beclomethasone or fluticasone treatment followed by a 4 week study drug washout with resumption of standard asthma medication regimen for 4 weeks, followed by 8 weeks of beclomethasone or fluticasone (whichever drug was not taken the first 8 weeks)
  Interventions: Drug: beclomethasone
- fluticasone (Experimental): Subjects are being randomized to 8 weeks of beclomethasone or fluticasone treatment followed by a 4 week study drug washout with resumption of standard asthma medication regimen for 4 weeks, followed by 8 weeks of beclomethasone or fluticasone (whichever drug was not taken the first 8 weeks)
  Interventions: Drug: fluticasone

INTERVENTIONS:
Drug: beclomethasone
  Arms: Beclomethasone
Drug: fluticasone
  Arms: fluticasone

SUMMARY:
The primary objective of the study is to show that ventilation heterogeneity identified by hyperpolarized helium-3 lung MRI is prevalent children with poorly controlled asthma despite guidelines-based treatment with ICS. The secondary objective is to demonstrate whether or not eight weeks of treatment with extra-fine particle ICS (HFA-BDP) improves ventilation heterogeneity compared to treatment with a coarse particle ICS (fluticasone HFA or dry powder).

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls between the ages of 6 and 17 years
* Diagnosis of asthma based on NAEPP3 criteria
* Poor asthma control based on one or more of the following criteria:

an ACT ≤ 19 and/or ACQ ≥ 1.5 units at the screening and/or randomization visits despite continuous or intermittent treatment with ICS and/or an anti-leukotriene within six months before enrollment.

* Any airflow obstruction based on Hankinson et al reference standards: FEV1 % < 80% predicted, an FEV1/FVC ratio < 90% predicted, and/or an FEF 25-75 < 70% predicted at the screening and/or randomization visits.
* Frequent severe exacerbations as reflected by ≥ 2 bursts of systemic corticosteroids (≥ 3 days each) in the previous 12 months.
* Serious exacerbations reflected by at least one hospitalization, ICU stay, or mechanical ventilation in the previous 12 months
* "Not well controlled" by NAEPP or GINA asthma treatment guidelines
* For post-pubertal females, negative urine pregnancy screen and willing if sexually active (as counseled by a female study coordinator in private) to using a consistent and appropriate method of birth control for the duration of the study.

Exclusion Criteria:

* Premature birth < 35 weeks estimated gestational age
* Maintenance oral prednisone (defined as daily or alternate day for the past three months before screening) or omalizumab treatment for asthma control
* Any significant medical condition that might inform maldistribution of ventilation apart from asthma including bronchiectasis, cardiac disease, congenital anomalies of the respiratory system, neurodevelopmental delay with cognitive impairment, ciliary dyskinesia syndromes, immune deficiency, recent lower respiratory infection (within six weeks of screen visit). Co-morbidities associated with asthma including sleep apnea syndrome, obesity, GERD, and right middle lobe syndrome are not criteria for exclusion.
* Claustrophobia, inner ear implants, aneurysm or other surgical clips, metal foreign bodies in the eye, pacemaker, or other contraindication to MR scanning. Subjects with any implanted device that cannot be verified as MRI compliant will be excluded.
* Chest circumference greater than that of the helium coil. The circumference of the coil is approximately 42 inches.
* Inability to understand simple instructions or to hold still for 10 seconds.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Ventilation Heterogeneity Index (VHI) | Baseline
  VHI = lung defect volume divided by total lung volume. It is a ratio scale.

SECONDARY OUTCOMES:
Change in Ventilation Heterogenity Index (VHI) | Baseline (week 0), week 12, week 16, and week 24
  VHI = lung defect volume divided by total lung volume. This is a ratio scale that will be measured at four timepoints: enrollment (week 0), end of treatment 1(week 12), start of treatment 2 (week 16), and end of treatment 2 (week 24). The VHI will be compared at the beginning and end of phase 1 and at the beginning and end of phase two using ANOVA based on a mixed-effects model, with fixed effects of sequence, period, and treatment of a random effect of subject within sequence, and baseline covariate.

CONTACTS AND LOCATIONS:
Overall Officials: W. Gerald Teague, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia - Fontaine Research Park, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Gerald Teague W, Mata J, Qing K, Tustison NJ, Mugler JP, Meyer CH, de Lange EE, Shim YM, Wavell K, Altes TA. Measures of ventilation heterogeneity mapped with hyperpolarized helium-3 MRI demonstrate a T2-high phenotype in asthma. Pediatr Pulmonol. 2021 Jun;56(6):1440-1448. doi: 10.1002/ppul.25303. Epub 2021 Feb 23. PMID 33621442